CLINICAL TRIAL: NCT02365818
Title: An Open Label, Single Arm, Phase II, Multicenter Study of the Safety and Efficacy of CG0070 Oncolytic Vector Regimen in Patients With Non-Muscle Invasive Bladder Carcinoma Who Have Failed BCG (Bacillus Calmette-Guerin) Therapy and Refused Cystectomy
Brief Title: Safety and Efficacy of CG0070 Oncolytic Virus Regimen for High Grade NMIBC After BCG Failure
Acronym: BOND2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CG Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOND 2 version 3.8
Record Dates: First submitted 2015-02-09; First posted 2015-02-19 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CG0070 (Experimental): Single arm intervention with CG0070 to be given at a dose of 1e12 vp weekly for six weeks. Patients who achieve a partial response or a complete response at 6 months post first intravesical intervention will be maintained with the same induction cycle of weekly times six. Patients will be followed every 3 months through Month 24.
  Interventions: Biological: CG0070

INTERVENTIONS:
Biological: CG0070
  Other Names: oncolytic adenovirus with a E2F promotor and expresses GMCSF

SUMMARY:
To study the safety and efficacy of CG0070, an oncolytic virus expression GM-CSF in high grade non muscle invasive bladder cancer patients who failed BCG therapy and refused cystectomy.

DETAILED DESCRIPTION:
The plan is to study the safety and efficacy of CG0070 in high-grade NMIBC (Non-muscle Invasive Bladder Cancer) patients who failed BCG therapy. Most patients with NMIBCis (Cis, Cis with Ta and/or T1, high grade Ta or T1 with frequent or uncontrolled recurrences) who have failed BCG (Bacillus Calmette-Guerin) intravesical therapy (standard of care) usually have no other choice but to proceed to cystectomy. Cystectomy is a surgery associated with major morbidity, mortality and quality of life issues. Morbidity and long term tedious medical care will be for the rest of the patient's life span. Most patients at this stage do not show signs of disease progression into the muscle layer or of metastasis, making surgery a very difficult decision. CG0070, if successful in this trial, will serve to provide a therapeutic alternative for this patient population in need.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically confirmed non-muscle invasive bladder cancer (NMIBC) high grade disease (HG), as defined by the 2004 WHO classification system
2. Patients must have no evidence of muscle invasive disease
3. Patients must be able to provide a sufficient biopsy sample to the central pathologist for histopathologically confirmed, transitional cell (urothelial) carcinoma. Urothelial tumors with mixed histology (but with <50% variant) are eligible.
4. Patients must have received at least two or more prior courses of intravesical therapy per recommended schedules. Bacillus Calmette-Guerin (BCG) must have been one of the prior therapies administered.
5. Patients can have either failed BCG induction therapy within a six-month period or have been successfully treated with BCG, but subsequently found to have recurrence. The first standard course of intravesical BCG therapy must include at least six weekly treatments (allowable range of instillations per course is 4-9). The second course of BCG therapy must include at least two weekly treatments.
6. Patients have either Cis or Cis with Ta and/or T1 disease at enrollment or in the past. For those patients with only Ta or T1 disease at enrollment AND with no history of Cis, they must have

   * disease recurrence either must occur within 12 months of the most recent intravesical therapy of any kind, OR
   * disease recurrence within 18 months of BCG maintenance OR
   * disease recurrence within 24 months of BCG induction
   * T1 patients need to have evidence of muscle included in their latest biopsy; and if not a re-TURBT has to be done prior to enrollment
7. 18 years of age or older
8. Radical cystectomy has been declined by the patient in a signed special section of the informed consent, whereby there is a clear explanation by the investigator to the subject that a delay of cystectomy may increase his/her chance of disease progression, the results of which may lead to serious and life threatening consequences.
9. Patients must be able to enter into the study within ten weeks of their most recent diagnostic procedure, which is usually a diagnostic biopsy, a transurethral resection of bladder tumor (TURBT) procedure or positive urine cytology.
10. Eastern Cooperative Oncology Group (ECOG) performance status <2.
11. Not pregnant or lactating
12. Patients with child bearing potential must agree to use adequate contraception
13. Agree to study specific informed consent and HIPAA authorization for release of personal health information
14. Adequate baseline CBC, renal and hepatic function. Parameters described as WBC>3000 cells/mm^3, ANC>1,000 cells/mm^3, hemoglobin>9.5g/dL, and platelet count >100,000 cells/mm^3

    * Adequate renal function: serum creatinine <2.5mg/dL
    * Bilirubin, AST and ALT not more than 2 x Upper Limits of Normal
    * PT/INR, PTT, and fibrinogen within institutional acceptable limits
    * Absolute lymphocyte count ≥ 800/μL before the first dose of CG0070

Exclusion Criteria:

1. Previous systemic chemotherapy or radiation for bladder cancer. Note: Prior immunotherapy or intravesical (administered within the bladder) chemotherapy for superficial disease is acceptable
2. History of anaphylactic reaction following exposure to humanized or human therapeutic monoclonal antibodies, hypersensitivity to GM-CSF or yeast derived products, clinically meaningful allergic reactions or any known hypersensitivity or prior reaction to any of the formulation excipients in the study drugs.
3. Known infection with HIV, HBV or HCV.
4. Anticipated use of chemotherapy or radiotherapy not specified in the study protocol while on study
5. Any underlying medical condition that, in the Investigator's opinion, will make the administration of study vector hazardous to the patient, would obscure the interpretation of adverse events, or not permit adequate surgical resection.
6. Systemic treatment on any investigational clinical trial within 28 days prior to registration.
7. Concurrent treatment with immunosuppressive or immunomodulatory agents, including any systemic steroid (exception: inhaled or topically applied steroids, and acute and chronic standard dose NSAIDs, are permitted). Use of a short course (i.e., ≤ 1 day) of a glucocorticoid is acceptable to prevent a reaction to the IV contrast used for CT scans.
8. Immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 3 months of study entry.
9. History of prior experimental cancer vaccine treatment (e.g., dendritic cell therapy, heat shock vaccine) within the last year
10. History of stage III or greater cancer, excluding urothelial cancer. Basal or squamous cell skin cancers must have been adequately treated and the subject must be disease-free at the time of registration. Subjects with a history of stage I or II cancer, must have been adequately treated and have been disease-free for ≥ 2 years at the time of registration.
11. Progressive or persistent viral or bacterial infection

    * All infections must be resolved and the patient must remain afebrile for seven days without antibiotics prior to being placed on study
    * Urinary tract infection, including particularly bladder infection, must be resolved prior to being placed on study
12. Unwilling or unable to comply with the protocol or cooperate fully with the investigator and site personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Durable Complete Response Proportion (DCR) | 18 months time point from the date of the first intravesical intervention
  Defined as the proportion of patients who experience a durable complete response lasting 12 months or longer from the initial confirmed complete response date (first CR assessment to be at least 6 months after the first intravesical intervention) and at least 18 months from the date of the first intravesical intervention

SECONDARY OUTCOMES:
Cystectomy Free Survival | 18 months after the first intravesical treatment
  Not available, not collected on study or not currently available
Complete Response Survival | 18 months after the first intravesical treatment
  Not available, not collected on study or not currently available
Progression Free Survival | 18 months after the first intravesical treatment
  Not available, not collected on study or not currently available
Time to Progression to Muscle Invasive Disease | 18 months after the first intravesical treatment
  Not available, not collected on study or not currently available
Overall Survival | 18 months and 24 months after first intravesical treatment
  Not available, not collected on study or not currently available
PD-L1 Status Changes | changes between pre-intervention and post intervention at either cystectomy or at biopsy up to 24 months
  PD-L1 status of cancer cells and immune cells at tumor site by IHC
Organ Confined Disease Proportions | at cystectomy
  Patient proportions with no cancer cells in regional lymph nodes at cystectomy
Complete Response Proportions | 24 months after the first intravesical treatment
  Proportions of patients with a complete response of at least 12 months' duration
PD-1 Status Changes | changes between pre-intervention and post intervention at either cystectomy or at biopsy up to 24 months
  PD-1 status of immune cells at tumor site by IHC
Disease Regression Proportions | 24 months after the first intravesical treatment
  Proportions of patients with a partial response and/or a complete response of less than 12 months' duration

CONTACTS AND LOCATIONS:
Overall Officials: Gary Steinberg, MD, Principal Investigator — University of Chicago
Locations (17):
- United States (17):
  - Alaska Clinical Research Center, Anchorage, Alaska
  - BCG Oncology, Phoenix, Arizona
  - Arizona Institute of Urology, Tucson, Arizona
  - Institute of Urologic Oncology at UCLA, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - University of California, San Diego, San Diego, California
  - UF Health Cancer Center, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Michigan Institute of Urology, P.C., Troy, Michigan
  - Adult Pediatric Urology and Urogynecology, PC, Omaha, Nebraska
  - GU Research Network/ The Urology Center, Omaha, Nebraska
  - Premier Urology Group, LLC., Edison, New Jersey
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Dept. of Urologic Surgery, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin